CLINICAL TRIAL: NCT06574152
Title: Effect of Photobiomodulation on Pain and Healing of the Vertical Releasing Incision After Endodontic Microsurgery: A Randomized Clinical Trial
Brief Title: Effect of Photobiomodulation on Pain and Healing of the Vertical Releasing Incision After Endodontic Microsurgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Juliana Barros, DDS, MS, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-24-0527
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Apical Periodontitis; Endodontically Treated Teeth; Endodontic Disease; Apical Cyst; Apical Granuloma; Periradicular Disease; Previous Endodontic Treatment
Keywords: vertical incision; photobiomodulation; apicoectomy; endodontic microsurgery; laser therapy
MeSH Terms: conditions — Periapical Periodontitis; Tooth, Nonvital; Dental Pulp Diseases; Radicular Cyst; Periapical Granuloma; Periapical Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EMS and PBM treatment (Experimental): Photobiomodulation (PBM) therapy will be performed using a 660 nm diode laser (SiroLaser Advance Plus, Dentsply Sirona Inc, Charlotte, North Carolina, USA) following the outline of the incision flap in a contact mode. Each site will be irradiated for 25 seconds with an energy density of 10 J/cm2 (irradiation mode).
  Interventions: Device: PBM treatment; Device: EMS
- EMS and PBM sham treatment (Sham Comparator): The laser tip will be placed following the outline of the incision flap in a contact mode but without activating it (no irradiation).
  Interventions: Device: PBM sham treatment; Device: EMS

INTERVENTIONS:
Device: PBM treatment — Immediately after the apical microsurgery, PBM therapy will be performed using a 660 nm diode laser (SiroLaser Advance Plus, Dentsply Sirona Inc, Charlotte, North Carolina, USA), with an 8 mm tip diameter . The laser tip will be placed following the outline of the incision flap in a contact mode . The power output of the laser will be 50 milliwatt (mW) and verified by a Power Meter (PM600 Power/Energy meter, Molectron Detector Inc, Portland, OR, USA). Each site will be irradiated for 25 s with an energy density of 10 J/cm2
  Arms: EMS and PBM treatment
Device: PBM sham treatment — Immediately after the apical microsurgery, sham therapy will be performed without activating the laser.
  Arms: EMS and PBM sham treatment
Device: EMS — Patients will be anesthetized. All surgeries will be performed using a surgical microscope. After reflection of a mucoperiosteal flap, osteotomies will be performed to access the root apices and apical lesions. Root apices will be resected at 3 mm, and the pathological tissue curetted out. Next, root-end preparations will be made with ultrasonic tips and filled with calcium silicate-based materials. Methylene blue dye will be used for inspection after root-end resection before the root-end preparation and filling. After cleaning the osseous crypt, the wound margins will be reapproximated with 5-0 single interrupted sutures. A gauze will be placed for 30 minutes for wound compression. Sutures will be removed seven days postoperatively

SUMMARY:
The purpose of this study is to evaluate the effect of Photobiomodulation (PBM) in postoperative pain after endodontic microsurgery (EMS) in patients from the University of Texas Health Science Center at Houston, School of Dentistry Graduate Endodontic Clinic and to assess the soft tissue healing of the vertical releasing incision (VRI) after PBM

DETAILED DESCRIPTION:
From the University of Texas Health Science Center School of Dentistry at Houston (UTHealth), forty patients needing endodontic microsurgery (EMS) (where the tissue flap design includes vertical releasing incisions) will be recruited for this study.

Photobiomodulation (PBM) has been used for decades in medicine and dentistry showing promising results in the healing capabilities, however, an accepted protocol has still not been created for its regular use in endodontics. PBM functions on the principle of harnessing light energy to stimulate cellular activity, particularly with the mitochondria (Karu, 2008). When specific wavelengths of light, typically in the red or near-infrared spectrum, penetrate the tissue, a series of photochemical reactions occur. This light energy enhances the production of adenosine triphosphate (ATP), the primary source of cellular energy, leading to improved cellular function and metabolism. Additionally, photobiomodulation can influence various cellular processes, such as reducing oxidative stress and inflammation, ultimately promoting less postoperative pain and enhanced soft tissue healing (Sobouti et al., 2015, Fulop et al., 2010, Sanz-Moliner et al., 2013).

Findings regarding the quality of life after apical surgery suggest that patients commonly hold negative beliefs and perceive it as one of the most painful among endodontic procedures (Morse et al., 1990), when in fact, it could be less unpleasant than expected (Iqbal et al., 2007). Apical surgery has significantly evolved with the introduction of the surgical operating microscope and microsurgical instruments, transforming it into a distinct and more successful procedure. The adoption of microsurgical techniques has been associated with reduced postoperative pain (Pecora et al., 1993), likely due to minimized tissue trauma and enhanced precision facilitated by superior visualization.

Consequently, since PBM can promote pain relief, tissue repair, and regeneration, it may serve as a valuable tool for EMS, reducing postoperative pain and improving overall healing (Mizutani et al., 2016).

Forty adult patients will be invited to participate in this study. They will be divided into two groups: (A) Experimental group (n=20) where patients will receive conventional EMS and PBM treatment, and (B) Control group (n=20) where patients will receive conventional EMS and PBM sham treatment. Preoperative and postoperative pain will be assessed using a visual analog pain scale and the tissue healing will be evaluated by visual inspection and photographs.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I or II.
* At least one tooth will receive EMS.
* Flap design that includes at least one VRI (triangular, rectangular, papilla base or submarginal rectangular).

Exclusion Criteria:

* ASA III or IV.
* Current heavy smokers (>10 cigarettes/day)
* Uncontrolled diabetes (HbA1c ≥ 7%) or other uncontrolled systemic diseases that may comprise healing, such as vitamin C deficiency, neutrophil deficiencies, immunodeficiency syndromes, or leukemia.
* Surgical access on the palatal surface.
* Acute swelling or abscess present on the day of the surgery.
* Any event or condition that would make continued participation in the study not in the best interest of the subject, as determined by the investigator.
* Pregnancy.
* Development of any medical condition that might affect the treatment and clinical outcomes, as determined by the investigator.
* Initiation of any treatment or exposure that might affect therapy's healing, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain as assessed by a Visual Analogue Scale (VAS) | preoperative assessment (baseline), in the day of the intervention (surgery day) and 5-7 days after the surgery (sutures removal appointment).
  this is scored on a likert scale from 0(no pain), 1-3(mild pain), 4-6( moderate pain to 10(worst pain)

SECONDARY OUTCOMES:
Change in healing as assessed by the Early Wound Healing Score (EHS). | preoperative assessment (baseline), immediately after surgery, and 5-7 days post-surgery during the sutures removal appointment
  The EHS is composed of 3 parameters: clinical signs of re-epithelization (CSR), clinical signs of hemostasis (CSH), and clinical signs of inflammation (CSI).
  Zero (visible distance between incision margins), 3 (incision margins in contact), or 6(merged incision margins) points were used to evaluate CSR, whereas 0 (bleeding at the incision margins), 1 (presence of fibrin at the incision margins), or 2(absence of fibrin on the incision margins) points were used for CSH and 0 points (redness involving >50% of the incision length and/or pronounced swelling) 1 point (redness involving <50% of the incision length) 2 points (absence of redness along the incision length) were used to analyze CSI
  The summation of the points of these 3 parameters generated the EHS. The EHS for ideal wound healing was 10 points, while the worst possible score was 0 points

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Barros, DDS,MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No